CLINICAL TRIAL: NCT04901923
Title: A Phase 1, Single-center, Open-label, Sequential Dose-Escalation Study of ACP-196 in Healthy Subjects to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, Food Effects, and Drug-Drug Interactions
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, Food Effects, and Drug-drug Interactions of ACP-196 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-001
Record Dates: First submitted 2021-05-06; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Healthy Participants
Keywords: Acalabrutinib; ACP-196; Drug-drug interaction; Food effects; Healthy participants; Itraconazole; Pharmacodynamics; Pharmacokinetics; PK
MeSH Terms: interventions — acalabrutinib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Cohort 1 (Experimental): Participants will receive ACP-196 2.5 mg capsule orally BID on Day 1.
  Interventions: Drug: ACP-196
- Part 1 Cohort 2 (Experimental): Participants will receive ACP-196 5 mg (2 x 2.5 mg capsules) orally BID on Day 1.
  Interventions: Drug: ACP-196
- Part 1 Cohort 3 (Experimental): Participants will receive ACP-196 25 mg capsule orally BID on Day 1.
  Interventions: Drug: ACP-196
- Part 1 Cohort 4 (Experimental): Participants will receive ACP-196 50 mg (2 x 25 mg capsules) orally BID on Day 1.
  Interventions: Drug: ACP-196
- Part 1 Cohort 5 (Experimental): Participants will receive ACP-196 100 mg (4 x 25 mg capsules) orally QD on Day 1.
  Interventions: Drug: ACP-196
- Part 2 Cohort 6 (Experimental): Participants will receive ACP-196 75 mg (3 x 25 mg capsules) orally QD on Day 1 and Day 8.
  Interventions: Drug: ACP-196
- Part 3 Cohort 7 (Experimental): Participants will receive ACP-196 50 mg (2 x 25 mg capsules) orally QD on Day 1, itraconazole 200 mg capsules BID from Days 4 to 8 with meals and then ACP-196 50 mg (2 x 25 mg capsules) along with itraconazole 200 mg capsule QD on Day 9 under fasting state.
  Interventions: Drug: ACP-196; Drug: Itraconazole

INTERVENTIONS:
Drug: ACP-196 — Participants will receive ACP-196 oral capsule(s) in all parts.
  Other Names: Acalabrutinib
Drug: Itraconazole — Participants will receive itraconazole 200 mg capsules BID from Days 4 to 8 with meals and then 200 mg capsule QD on Day 9 under fasting state.
  Arms: Part 3 Cohort 7

SUMMARY:
This study is to evaluate the safety, pharmacokinetics/pharmacodynamics (PK/PD), food-effect, and drug-drug interaction study of ACP-196 in healthy participants.

DETAILED DESCRIPTION:
The study is divided into 3 parts. Part 1 will include 5 cohorts (Cohorts [C] 1 to 5) and participants will receive oral ACP-196 2.5 to 50 mg twice daily (BID) and 100 mg once daily (QD) on Day 1. In Part 2 (Cohort 6), participants will receive a single oral dose of 75.0 mg QD in a fasting and a fed state, with a 7-day washout period between the 2 doses. In Part 3 (Cohort 7), participants will receive a single oral dose of 50.0 mg QD alone on Day 1 and in combination with itraconazole on Day 9. Itraconazole 200 mg will be given twice daily (12 hours apart) with meals on Days 4 to 8 and once on Day 9 with ACP-196 under a fasting state in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >=18.0 and <=30.0 kg/m^2.
* Healthy as determined by medical history and physical examination.
* Nonsmoker
* Normal clinical laboratory test results and ECG, or results with minor deviations which are not considered to be clinically significant in the judgment of the investigator.
* Men of and women of childbearing potential to follow protocol defined contraception methods.
* Women must have negative urine pregnancy test.
* Willingness and ability to swallow study drug capsules.

Exclusion Criteria:

* Prior or ongoing clinically significant illness, medical condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject; alter the absorption, distribution, metabolism, or excretion of the study drug; or impair the assessment of study results.
* Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections).
* Women cannot be pregnant or breast feeding.
* Significant history of drug or alcohol abuse or addiction within 3 years before study screening or as evidenced by continuing medical complications of prior drug or alcohol use.
* History of blood or plasma donation within 90 days before first study drug administration.
* Currently drinking over 21 units/week of ethanol
* Drug toxicology screen positive for any prohibited drugs, illicit substances, or alcohol.
* Anticipated need for alcohol, tobacco, or any drug during the study drug administration and immediate follow-up periods.
* Relative to admission has any of the following exposures: has taken a prescription systemic medication within 14 days; has used an over-the counter systemic medication (other than acetaminophen) within 7 days; has ingested calcium supplements or calcium-containing vitamins within 7 days; has ingested grapefruit, grapefruit juice, or grapefruit-containing products within 7 days; has consumed alcohol within 48 hours; has taken acetaminophen within 24 hours.
* Positive test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen or hepatitis B core antibody, or hepatitis C antibody.
* Unwillingness to avoid vigorous physical activity during inpatient clinic confinements.
* Part 2 only - Inability or unwillingness to eat all of the ingredients of the high-fat, high-calorie meal as specified in the protocol.
* Part 3 only - Known allergy to itraconazole or other azole compounds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2014-05-22 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Maximum Observed Plasma Concentration (Cmax) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Time to reach Cmax (Tmax) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Terminal-elimination Half-life (T1/2) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Terminal-elimination Rate Constant (λz) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Time Delay Between the Time of Dosing and the First Measurable Concentration (tlag) of ACP-196 in Parts 1, 2, and 3 | Part 1: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 13, 14, 15, 16, 18, 20, 24, 36, 48, 60h; Parts 2 and 3: predose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72h; and till 48h on Day 8 of Part 2; and till 24h on Day 9 of Part 3
Incidences of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Part 1: Day 1 through Day 3; Part 2 and Part 3: Day 1 through Day 10
Incidences of Abnormal Vital Signs Reported as TEAEs | Part 1: Day 1 ( from 1 hr predose through 1 hr postdose); Part 2: From Day 1 (1 hr predose) through Day 8 (1 hr postdose); Part 3: From Day 1 (1 hr predose) through Day 9 (1 hr postdose)
Incidences of Abnormal Clinical Laboratory Parameters Reported as TEAEs | Part 1: From Day 1 to Day 2; Part 2 and Part 3: From Day 1 to Day 10
Incidences of Abnormal Electrocardiograms (ECGs) Reported as TEAEs | Part 1: Day 1 ( from 1 hr predose through 1 hr postdose); Part 2: From Day 1 (1 hr predose) through Day 8 (1 hr postdose); Part 3: From Day 1 (1 hr predose) through Day 9 (1 hr postdose)

SECONDARY OUTCOMES:
Occupancy of Bruton's Tyrosine Kinase (BTK) by ACP-196 in Peripheral Blood Mononuclear Cells (PBMCs) | 1, 3, 12, 15, and 24 hrs after first dose on Day 1
  The BTK occupancy will be measured by BTK occupancy assay which measures percent of BTK occupied post baseline compared to the baseline, post administration of study drug. The BTK occupancy is defined as ACP-196 active-site occupancy of > 80% at 24 hours after the first dose administration.
Effect of ACP-196 on Biologic Markers of B-cell Function | 1, 3, 12, 15, and 24 hrs after first dose on Day 1
  The pharmacodynamics of ACP-196 will be evaluated in cluster of differentiation (CD) 69/CD86 expression. It will be considered as complete inhibition when biological markers of B-cell function (CD69 and CD86) inhibition ≥ 90%.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home